CLINICAL TRIAL: NCT01712334
Title: A Phase IV Multicenter, Randomized, Open Label, Two-Period, Crossover Study in Patients With Cystic Fibrosis to Evaluate the Comparable Efficacy and Safety of Pulmozyme Delivered by the eRapid Nebulizer System
Brief Title: A Study of the Comparable Efficacy and Safety of Pulmozyme (Dornase Alfa) Delivered by the eRapid Nebulizer System in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML28249
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — dornase alfa

ARMS (2):
- eRapid Nebulizer (Experimental): Dornase alfa (Pulmozyme®) inhaled once daily by the Pari eRapid nebulizer for 2 weeks.
  Interventions: Drug: dornase alfa [Pulmozyme®]
- Jet Nebulizer (Active Comparator): Dornase alfa (Pulmozyme®) inhaled once daily by the Pari LC Plus jet nebulizer for 2 weeks.
  Interventions: Drug: dornase alfa [Pulmozyme®]

INTERVENTIONS:
Drug: dornase alfa [Pulmozyme®] — Inhaled once daily by Pari eRapid nebulizer.
  Arms: eRapid Nebulizer
Drug: dornase alfa [Pulmozyme®] — Inhaled once daily by Pari LC Plus jet nebulizer.
  Arms: Jet Nebulizer

SUMMARY:
This phase IV, multicenter, randomized, open-label, two-period crossover study will evaluate the comparable efficacy and safety of Pulmozyme (dornase alfa) delivered by the eRapid nebulizer system in patients with cystic fibrosis. Patients who have been receiving Pulmozyme once daily chronically for at least 6 months will continue to receive Pulmozyme once daily for a run-in period of 2 weeks using the Pari LC Plus nebulizer. Patients will then be randomized to receive in a crossover design Pulmozyme once daily for two treatment periods of 2 weeks each using either the Pari LC Plus or the eRapid nebulizer. Anticipated time on study treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, >/= 6 years of age
* Confirmed diagnosis of cystic fibrosis (CF)
* Receiving Pulmozyme once daily chronically for treatment of CF for at least 6 months prior to screening
* Percent predicted FEV1 >/= 40% at screening based on the Wang (males < 18 years, females < 16 years) or Hankinson (males >/= 18 years, females >/= 16 years) standardized equations
* Able to reproducibly perform spirometry testing and comply with study assessments

Exclusion Criteria:

* An acute respiratory infection or pulmonary exacerbation within 4 weeks prior to randomization
* Initiation of any new chronic therapy (e.g. inhaled corticosteroids, inhaled oral antibiotics, high-dose ibuprofen, hypertonic saline, ivacaftor) for respiratory disease within 4 weeks prior to randomization
* Changes in chest physiotherapy schedule within 4 weeks prior to randomization
* Hospitalization within 4 weeks prior to randomization
* Planned hospitalization during the 6-week study
* History of organ transplantation
* Participation in an investigational drug or device study within 30 day prior to screening

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (16):
- United States (16):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Portland, Maine
  - Boston, Massachusetts
  - Lebanon, New Hampshire
  - Long Branch, New Jersey
  - Rochester, New York
  - Durham, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Nashville, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington

REFERENCES:
- [Derived] Yang C, Montgomery M. Dornase alfa for cystic fibrosis. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD001127. doi: 10.1002/14651858.CD001127.pub5. PMID 33735508
- [Derived] Sawicki GS, Chou W, Raimundo K, Trzaskoma B, Konstan MW. Randomized trial of efficacy and safety of dornase alfa delivered by eRapid nebulizer in cystic fibrosis patients. J Cyst Fibros. 2015 Nov;14(6):777-83. doi: 10.1016/j.jcf.2015.04.003. Epub 2015 Apr 25. PMID 25921451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 99 patients were enrolled. 96 unique patients entered the run-in period including 3 patients who entered the run-in period twice.
Pre-assignment Details: Patients received dornase alfa (Pulmozyme®) by LC Plus nebulizer in the 2-week run-in period prior to randomization. A total of 86 unique patients were randomized in the study in 87 randomization events. Of the randomized patients, 85 patients completed the study in two treatment sequences.
Groups:
- eRapid Nebulizer Then Jet Nebulizer: Dornase alfa (Pulmozyme®) inhaled once daily by the Pari eRapid nebulizer for 2 weeks in Treatment Period 1 then Pulmozyme® inhaled once daily by the Pari LC Plus jet nebulizer for 2 weeks in Treatment Period 2.
  .
- Jet Nebulizer Then eRapid Nebulizer: Pulmozyme® inhaled once daily by the Pari LC Plus jet nebulizer for 2 weeks in Treatment Period 1 then Pulmozyme® inhaled once daily by the Pari eRapid nebulizer for 2 weeks in Treatment Period 2.
Period: Treatment Period 1
Arm/Group | eRapid Nebulizer Then Jet Nebulizer | Jet Nebulizer Then eRapid Nebulizer
Started | 44 | 43
Received Treatment | 44 | 41
Completed | 44 | 41
Not Completed | 0 | 2
Not completed — Randomized in Error | 0 | 2
Period: Treatment Period 2
Arm/Group | eRapid Nebulizer Then Jet Nebulizer | Jet Nebulizer Then eRapid Nebulizer
Started | 44 | 41
Completed | 44 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures were based on the modified Intent-to-Treat (mITT) population that included all participants randomized with both baseline and endpoint Forced Expiratory Volume in 1 second (FEV1) values for both treatment periods.
Groups:
- All Participants: All participants received dornase alfa (Pulmozyme) inhaled once daily by the Pari eRapid nebulizer or the Pari LC Plus jet nebulizer for 2 weeks in Treatment Period 1 then crossed over to use the other nebulizer in Treatment Period 2 for 2 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Stability of Lung Function: Percent Predicted Forced Expiratory Volume in 1 Second (FEV1)
Description: Spirometry was performed according to American Thoracic Society standards. FEV1 is the amount of air that is forced out of the lungs in one second and was measured at the end of each 2-week treatment period. The percent predicted FEV1 was calculated as: Percent predicted FEV1 =FEV1 (L) / Predicted FEV1 (L) ×100.
Time Frame: At the end of each 2-week treatment period
Population: Modified Intent-to-Treat (mITT) population included all randomized participants with baseline and endpoint FEV1 values for both treatment periods.
Measure: Mean (Standard Deviation); unit: percent predicted
Groups:
- Jet Nebulizer: Pulmozyme® inhaled once daily by the Pari LC Plus jet nebulizer for 2 weeks.
Arm/Group | eRapid Nebulizer | Jet Nebulizer
Number analyzed (Participants) | 85 | 85
percent predicted | 98.1 (22.1) | 97.2 (20.7)
Statistical Analysis 1: Comparison: eRapid Nebulizer vs Jet Nebulizer; Test type: Non-Inferiority or Equivalence — The ratio of the mean percent predicted FEV1 at the end of the eRapid treatment to the mean percent predicted FEV1 at the end of the LC Plus jet nebulizer treatment. The two nebulizers were considered equivalent if the 90% CI was within 80%-125%; Ratio (Fieller's theorem) = 100.9, 90% CI 2-sided [99.5 to 102.3]

2. Primary Outcome: Safety: Number of Participants With Adverse Events During Each Treatment Period
Description: An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study and laboratory or clinical tests that resulted in a change in treatment or discontinuation from study drug were reported as adverse events.
Time Frame: 4 Weeks
Population: Safety population included all randomized participants who received treatment.
Measure: Number; unit: participants
Arm/Group | eRapid Nebulizer | Jet Nebulizer
Number analyzed (Participants) | 85 | 85
participants | 18 | 24

ADVERSE EVENTS:
Description: Safety population included all randomized participants who received treatment.
Arm/Group | eRapid Nebulizer | Jet Nebulizer
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.